CLINICAL TRIAL: NCT01014520
Title: Comparative Effects of Single Dose Preemptive Gabapentin or Amitriptyline on Postoperative Pain and Opioid Consumption in Single Level Lumbar Laminectomy and Diskectomy: A Double Blind RCT With Placebo Control
Brief Title: Efficacy of Gabapentin or Amitriptyline to Reduce Postoperative Pain After Lumbar Laminectomy and Diskectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tabriz University (Other)
Responsible Party: Tabriz University, Tabriz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 883
Record Dates: First submitted 2009-11-14; First posted 2009-11-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Herniated Disc; Intervertebral Disc Displacement
Keywords: Lumbar; Diskectomy; Laminectomy
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Gabapentin; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): Neurontin
  Interventions: Drug: Gabapentin , Amitriptyline
- Amitriptyline (Experimental): Elavil
  Interventions: Drug: Gabapentin , Amitriptyline

INTERVENTIONS:
Drug: Gabapentin , Amitriptyline — Capsule, 300 mg, oral, single dose 2 hours before surgery
  Capsule,300 mg containing 25 mg Amitriptyline, oral, single dose 2 hours before surgery
  Other Names: Neurontin; Elavil

SUMMARY:
The hypothesis of this study is that Gabapentin or Amitriptyline has no role in preemptive analgesia to reduce postoperative pain after lumbar diskectomies.

DETAILED DESCRIPTION:
Pain suppression plays a decisive role in patients' satisfaction following lumbar diskectomies, as the psychological component of the pain is a major cause of treatment failure.

Controversy exists whether preemptive prescription of gabapentin, as a known contributor to reduce postoperative pain, has a role in patients undergoing laminectomy for lumbar diskectomy or spinal canal stenosis.The aim of this study is to test the efficacy of amitriptyline and gabapentin in this group of neurosurgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Age:18 to 60
* Weight: 60 to 80 Kg
* ASA Class: I,II
* Concordant physical and imaging findings in favor of symptomatic lumbar disk herniation
* Single level lumbar disk herniation unresponsive to medical treatment

Exclusion Criteria:

* Previous consumption of Gabapentin or Amitriptyline
* Known allergy to investigated drugs
* Reluctant to sign informed consent
* Previous history of intolerance to narcotics
* Simultaneous lumbar diskectomy and a fusion technique
* Known renal failure
* Pregnancy
* Contraindications to Amitriptyline or Gabapentin prescription
* Unable to use PCA
* Habitual use of alcohol or opium
* History of analgesic consumption during the last 24hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
30% reduction in opium consumption in either study arms compared to the placebo group | Within the first 24 hours after surgery

SECONDARY OUTCOMES:
30% reduction in pain according to visual analogue scale in either study arms compared to the placebo group | Within the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Aghamohammadi, MD, Study Chair — Tabriz University; Payman Vahedi, MD, Principal Investigator — Tabriz University
Locations (1):
- Tabriz University of Medical Sciences, Tabriz, East Azerbayjan, Iran